CLINICAL TRIAL: NCT05371210
Title: SAIF: An End-to-end System for Assessment and Intervention of Frailty
Brief Title: An End-to-end System for Assessment and Intervention of Frailty
Acronym: SAIF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tan Tock Seng Hospital (Other)
Collaborators: Nanyang Technological University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2020/01163
Record Dates: First submitted 2022-05-05; First posted 2022-05-12 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2022-08

CONDITIONS: Frailty
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SAIF (Experimental): After completion of baseline assessment, participants were required to interact with the SAIF system for 4 months. They were followed up at 2-month (mid-way of intervention), 4-month (end of intervention), and 7-month (3 months post-intervention).
  Interventions: Other: SAIF
- Control (No Intervention): Participants received a one-time health pamphlet after completing baseline assessment. They were followed up at 2-month, 4-month and 7-month thereafter.

INTERVENTIONS:
Other: SAIF — Participants interacted with SAIF system at least 2-3 times per week; each session took up to 20 minutes.
  Arms: SAIF

SUMMARY:
The study aims to evaluate the feasibility and effectiveness of using SAIF (an end-to-end System for Assessment and Intervention of Frailty) to reduce the risk and delay the progress of physical frailty.

DETAILED DESCRIPTION:
SAIF is a personalised, community-based system for both assessment and intervention of frailty. It comprises of 8 modules categorised into

1. Interface: virtual nurse and caregiver gateway
2. Assessment: computerised screening using Fried Frailty Phenotype (FFP) and FRAIL instruments, Gamified Walking While Talking to assess frailty status and predictive analytics to predict participant's frailty risk
3. Intervention: Physical exercise kiosks (Cycling and Taichi) incorporated with games, polypharmacy management and nutrition recommendation

A total of 105 eligible community-dwelling older adults were recruited and randomised either to control arm or intervention arm using a single-consent Zelen's design. Allocation concealment was achieved using permutated block randomisation; both research assistant and participant were blinded to randomisation list during enrolment.

All participants completed baseline assessment and subsequent follow-up assessments (2-month, 4-month and 7-month). Additionally, participants in the intervention arm began SAIF interaction for a period of 4 months upon completion of their baseline assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Age 60 and above
2. CFS 4 or 5 / CFS 3 with FRAIL score at least 1 / CFS 3 with FPQ score at least 1
3. Ambulate for at least 10m without walking aid
4. English and/or Mandarin speaking

Exclusion Criteria:

1. Known diagnosis of dementia or CMMSE score <19
2. Parkinson's disease
3. Hip surgery within the last 6 months
4. Presence of end-stage organ failure, symptomatic heart conditions or COPD
5. Active arthritis
6. Hospitalisation within the last 1 month
7. Participants who are unable to provide consent

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2021-03-15 (Actual); Primary Completion 2022-06-16 (Actual); Study Completion 2022-06-16 (Actual)

PRIMARY OUTCOMES:
Change in frailty scores as measured by Fried Frailty Phenotype (FFP) | 4 months
  FFP consists of 5 physical criteria: exhaustion, slowness, weakness, weight loss and low physical activity. Total score of criteria classifies participants into 3 categories:
  Not Frail (score 0) Pre-frail (score 1-2) Frail (score 3-5)
Change in frailty scores as measured by Fried Frailty Phenotype (FFP) | 7 months
  FFP consists of 5 physical criteria: exhaustion, slowness, weakness, weight loss and low physical activity. Total score of criteria classifies participants into 3 categories:
  Not Frail (score 0) Pre-frail (score 1-2) Frail (score 3-5)
Change in physical performance scored based on Short Physical Performance Battery (SPPB) | 4 months
  SPPB is an assessment tool that evaluates function in older adults based on total score derived from measurement of gait speed, balance and chair stand tests. SPPB instrument has a score range of 0 (worst performance) to 12 (best performance).
Change in physical performance scored based on Short Physical Performance Battery (SPPB) | 7 months
  SPPB is an assessment tool that evaluates function in older adults based on total score derived from measurement of gait speed, balance and chair stand tests. SPPB instrument has a score range of 0 (worst performance) to 12 (best performance).
Correlation between SAIF system and Clinical Frailty Scale (CFS) for identification of pre-frailty and frailty | 4 months
  CFS is a 9-point validated clinical assessment tool to evaluate frailty and fitness of an older adult. Domains of scale includes functions, comorbidities and cognition. Score on scale can classify participant's fitness into categories: very fit (CFS 1), well (CFS 2), managing well (CFS 3), vulnerable (CFS 4), mildly frail (CFS 5), moderately frail (CFS 6), severely frail (CFS 7), severely frail (CFS 8) and terminally ill (CFS 9).
Correlation between SAIF system and Clinical Frailty Scale (CFS) for identification of pre-frailty and frailty | 7 months
  CFS is a 9-point validated clinical assessment tool to evaluate frailty and fitness of an older adult. Domains of scale includes functions, comorbidities and cognition. Score on scale can classify participant's fitness into categories: very fit (CFS 1), well (CFS 2), managing well (CFS 3), vulnerable (CFS 4), mildly frail (CFS 5), moderately frail (CFS 6), severely frail (CFS 7), severely frail (CFS 8) and terminally ill (CFS 9).

SECONDARY OUTCOMES:
Change in Health Education Impact Questionnaire (heiQ) scores | 4 months
  heiQ is a validated, self-reported instrument with 8 domains to comprehensively evaluate patient education program and self-management intervention. Each domain score ranges from 1 to 4; a higher score indicates better outcome.
Change in Health Education Impact Questionnaire (heiQ) scores | 7 months
  heiQ is a validated, self-reported instrument with 8 domains to comprehensively evaluate patient education program and self-management intervention. Each domain score ranges from 1 to 4; a higher score indicates better outcome.
Change in quality of life as measured by five-level version of the EuroQol five-dimensional questionnaire (EQ-5D-5L) | 4 months
  EQ-5D-5L is a validated, self-reported questionnaire that comprises 5 descriptive domains (mobility, self-care, usual activities, pain/discomfort and anxiety/depression) and self-rated health scale (0 being the worst health imagine and 100 being the best health imagine).
Change in quality of life as measured by five-level version of the EuroQol five-dimensional questionnaire (EQ-5D-5L) | 7 months
  EQ-5D-5L is a validated, self-reported questionnaire that comprises 5 descriptive domains (mobility, self-care, usual activities, pain/discomfort and anxiety/depression) and self-rated health scale (0 being the worst health imagine and 100 being the best health imagine).

CONTACTS AND LOCATIONS:
Overall Officials: Wee Shiong Lim, Principal Investigator — Tan Tock Seng Hospital
Locations (1):
- Tan Tock Seng Hospital, Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Borrat-Besson, C., Ryser, V.-A., amp; Wernli, B. (2013). Transition between frailty states - A European comparison. In A. Börsch-Supan, M. Brandt, H. Litwin, G. Weber (Eds.), Active ageing and solidarity between generations in Europe - First results from SHARE after the economic crisis, 175-186.
- [Background] Cesari M, Prince M, Thiyagarajan JA, De Carvalho IA, Bernabei R, Chan P, Gutierrez-Robledo LM, Michel JP, Morley JE, Ong P, Rodriguez Manas L, Sinclair A, Won CW, Beard J, Vellas B. Frailty: An Emerging Public Health Priority. J Am Med Dir Assoc. 2016 Mar 1;17(3):188-92. doi: 10.1016/j.jamda.2015.12.016. Epub 2016 Jan 21. PMID 26805753
- [Background] Chong MS, Tay L, Chan M, Lim WS, Ye R, Tan EK, Ding YY. Prospective longitudinal study of frailty transitions in a community-dwelling cohort of older adults with cognitive impairment. BMC Geriatr. 2015 Dec 29;15:175. doi: 10.1186/s12877-015-0174-1. PMID 26715536
- [Background] Dent E, Lien C, Lim WS, Wong WC, Wong CH, Ng TP, Woo J, Dong B, de la Vega S, Hua Poi PJ, Kamaruzzaman SBB, Won C, Chen LK, Rockwood K, Arai H, Rodriguez-Manas L, Cao L, Cesari M, Chan P, Leung E, Landi F, Fried LP, Morley JE, Vellas B, Flicker L. The Asia-Pacific Clinical Practice Guidelines for the Management of Frailty. J Am Med Dir Assoc. 2017 Jul 1;18(7):564-575. doi: 10.1016/j.jamda.2017.04.018. PMID 28648901
- [Background] Fairhall N, Langron C, Sherrington C, Lord SR, Kurrle SE, Lockwood K, Monaghan N, Aggar C, Gill L, Cameron ID. Treating frailty--a practical guide. BMC Med. 2011 Jul 6;9:83. doi: 10.1186/1741-7015-9-83. PMID 21733149
- [Background] Fried LP, Tangen CM, Walston J, Newman AB, Hirsch C, Gottdiener J, Seeman T, Tracy R, Kop WJ, Burke G, McBurnie MA; Cardiovascular Health Study Collaborative Research Group. Frailty in older adults: evidence for a phenotype. J Gerontol A Biol Sci Med Sci. 2001 Mar;56(3):M146-56. doi: 10.1093/gerona/56.3.m146. PMID 11253156
- [Background] Geraedts HA, Zijlstra W, Zhang W, Bulstra S, Stevens M. Adherence to and effectiveness of an individually tailored home-based exercise program for frail older adults, driven by mobility monitoring: design of a prospective cohort study. BMC Public Health. 2014 Jun 7;14:570. doi: 10.1186/1471-2458-14-570. PMID 24908049
- [Background] Gill TM, Gahbauer EA, Allore HG, Han L. Transitions between frailty states among community-living older persons. Arch Intern Med. 2006 Feb 27;166(4):418-23. doi: 10.1001/archinte.166.4.418. PMID 16505261
- [Background] Merchant RA, Chen MZ, Tan LWL, Lim MY, Ho HK, van Dam RM. Singapore Healthy Older People Everyday (HOPE) Study: Prevalence of Frailty and Associated Factors in Older Adults. J Am Med Dir Assoc. 2017 Aug 1;18(8):734.e9-734.e14. doi: 10.1016/j.jamda.2017.04.020. Epub 2017 Jun 13. PMID 28623152
- [Background] Mitnitski AB, Mogilner AJ, Rockwood K. Accumulation of deficits as a proxy measure of aging. ScientificWorldJournal. 2001 Aug 8;1:323-36. doi: 10.1100/tsw.2001.58. PMID 12806071
- [Background] Morley JE, Malmstrom TK, Miller DK. A simple frailty questionnaire (FRAIL) predicts outcomes in middle aged African Americans. J Nutr Health Aging. 2012 Jul;16(7):601-8. doi: 10.1007/s12603-012-0084-2. PMID 22836700
- [Background] Puts MTE, Toubasi S, Andrew MK, Ashe MC, Ploeg J, Atkinson E, Ayala AP, Roy A, Rodriguez Monforte M, Bergman H, McGilton K. Interventions to prevent or reduce the level of frailty in community-dwelling older adults: a scoping review of the literature and international policies. Age Ageing. 2017 May 1;46(3):383-392. doi: 10.1093/ageing/afw247. PMID 28064173
- [Background] Rockwood K, Song X, MacKnight C, Bergman H, Hogan DB, McDowell I, Mitnitski A. A global clinical measure of fitness and frailty in elderly people. CMAJ. 2005 Aug 30;173(5):489-95. doi: 10.1503/cmaj.050051. PMID 16129869
- [Background] Teo N, Gao Q, Nyunt MSZ, Wee SL, Ng TP. Social Frailty and Functional Disability: Findings From the Singapore Longitudinal Ageing Studies. J Am Med Dir Assoc. 2017 Jul 1;18(7):637.e13-637.e19. doi: 10.1016/j.jamda.2017.04.015. PMID 28648903
- [Background] Verghese J, Holtzer R, Lipton RB, Wang C. Mobility stress test approach to predicting frailty, disability, and mortality in high-functioning older adults. J Am Geriatr Soc. 2012 Oct;60(10):1901-5. doi: 10.1111/j.1532-5415.2012.04145.x. Epub 2012 Sep 24. PMID 23002714